CLINICAL TRIAL: NCT06711640
Title: A Pharmacokinetic, Safety, and Tolerability Study of LUCEMYRA in the Treatment of Opioid Withdrawal Management in Adolescent Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study withdrawn prior to enrollment due to strategic portfolio decisions following divestiture of the investigational product.
Sponsor: USWM, LLC (dba US WorldMeds) (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USWM-LX1-1014; 1UG3DA061620 (NIH)
Record Dates: First submitted 2024-11-19; First posted 2024-12-02 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Opioid Withdrawal (Disorder); Opioid Use Disorder
Keywords: Opioid Withdrawal Syndrome; LUCEMYRA; Lofexidine Hydrochloride; Opioid Withdrawal Management; Adolescent; opioid discontinuation; opioid; medications for opioid use disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — lofexidine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- LUCEMYRA: 0.54 mg (Experimental): The initial LUCEMYRA dose for this study will be based on weight. Participants who weigh ≥45 kg will receive three 0.18 mg tablets (0.54 mg) QID.
  Interventions: Drug: LUCEMYRA (lofexidine) tablets
- LUCEMYRA: 0.36 mg (Experimental): The initial LUCEMYRA dose for this study will be based on weight. Participants who weigh ≥30 to <45 kg will receive two 0.18 mg tablets (0.36 mg) QID.
  Interventions: Drug: LUCEMYRA (lofexidine) tablets

INTERVENTIONS:
Drug: LUCEMYRA (lofexidine) tablets — Tablets. Participants weighing ≥45 kg: three 0.18 mg tablets (0.54 mg) four times per day (QID). Participants weighing ≥30 to <45 kg: two 0.18 mg tablets (0.36 mg) QID.

SUMMARY:
The goal of this clinical study is to evaluate the pharmacokinetic (PK), safety, and tolerability of LUCEMYRA in adolescents age ≥12 to <18 years old abruptly discontinuing opioid use.

DETAILED DESCRIPTION:
This is a Phase 1, Open-label, PK, safety, and tolerability study of LUCEMYRA in adolescents aged ≥12 to <18 years abruptly discontinuing opioid use. The objectives of the study are to evaluate the PK parameters, as well as safety and tolerability. The effectiveness of LUCEMYRA on the signs and symptoms of acute opioid withdrawal will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Written minor assent obtained either in English or Spanish, as applicable, in accordance with local laws and Institutional Review Board (IRB) requirements. Additionally, written informed consent obtained from the participant's parent or LAR/guardian(s) in accordance with local laws and IRB requirements.
2. Participant is willing and able to comply with scheduled visits, study dosing, laboratory tests, and other study procedures.
3. Participant can swallow tablets the same size as LUCEMYRA.
4. Adolescent male or female participants ≥12 years and <18 years of age (at the time of study entry).
5. Minimum weight ≥30 kg.
6. Female participants of childbearing potential must agree to practice a medically acceptable method of contraception (e.g., intrauterine device, hormonal contraception started at least one full cycle before study enrollment or barrier method in conjunction with spermicide) for the duration of the study (including 2 months after study completion). With approval by the Investigator, participants' parents or legal guardians may select abstinence as a form of birth control if deemed more appropriate. For the purposes of this study, all females are considered of childbearing potential unless they are confirmed by the Investigator to be premenarchal, biologically sterile, or surgically sterile (e.g., hysterectomy, bilateral oophorectomy, tubal ligation).
7. All female participants, regardless of childbearing potential, must have a negative urine human chorionic gonadotropin (hCG) pregnancy test at Screening and prior to dosing on Day 1.
8. History of opiate use as confirmed by diagnosis of OUD according to the diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V); documentation of opioid use in the participant's medical record; or self-report of opioid use by participant and seeking treatment for OUD.
9. Reported use of fentanyl, heroin, morphine, or any opioid with a half-life similar to heroin or morphine such as Vicodin®, Lortab®, Lorcet®, Percocet®, Percodan®, Tylox®, or hydrocodone (by any route of administration), or oxycodone (oxycodone and oxycodone time-released formulation when crushed and snorted, injected, or swallowed after chewing) for at least 21 of the past 30 days and use within 2 days of admittance to the inpatient clinic.
10. Urine toxicology screen positive for opioids.
11. Vital signs measured in a seated position after the participant has rested for 5 minutes must be as follows:

    1. Heart rate: ≥60 beats per minute
    2. Systolic blood pressure: ≥100 mmHg
    3. Diastolic blood pressure: ≥65 mmHg

Exclusion Criteria:

1. Known or suspected pregnancy, planned pregnancy, or lactation.
2. Treatment with an investigational drug, device, or biological agent within 30 days prior to Screening, or during LUCEMYRA administration in this study.
3. Any medical illness, condition, or clinical finding that, in the opinion of the Investigator and/or the Sponsor, would put the participant at undue risk or interfere with the participant's ability to complete the study.
4. Any anticipated or scheduled surgery during the study period.
5. Major surgery within 30 days before Screening.
6. Have clinically significant abnormal laboratory values as determined by the Investigator.
7. Abnormal cardiovascular exam at Screening, including any of the following:

   1. Clinically significant abnormal ECG (e.g., second or third-degree heart block, uncontrolled arrhythmia)
   2. QT with Fridericia's correction (QTcF) of ≥450 msec
   3. History of QT interval prolongation Note: if the QTcF interval meets the above criteria, the value may be confirmed by repeating the measurement (twice, if necessary). If 2 of 3 values meet the above criteria, the participant will be excluded from participation.
8. Mild, moderate, or severe renal dysfunction, defined as an estimated glomerular filtration rate <90 mL/min/1.73 m2 at Screening.
9. Hepatic dysfunction as defined by either of the following:

   1. Aspartate aminotransferase or alanine aminotransferase >2 × upper limit of normal (ULN) at Screening; or
   2. Child-Pugh score of ≥7.
10. Metastatic cancer diagnosed within the previous year or diagnosis of any malignancy or neoplasm within 3 months prior to Screening, exclusive of basal cell carcinoma.
11. History of lack of tolerance or lack of response to LUCEMYRA.
12. Urine toxicology screen positive for methadone.
13. Self-reported use of methadone in the 14 days prior to Screening.
14. Current dependence, according to the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI KID) on any psychoactive substance (other than caffeine, nicotine, or the opioids listed in inclusion criterion #9) that requires detoxification or dose reduction as part of the pre-defined individual participant opioid withdrawal treatment goal.
15. A psychiatric disorder that, in the opinion of the Investigator, requires ongoing treatment making study participation unsafe or treatment compliance difficult.
16. History of suicidal behavior within the past 30 days or the participant is at risk of selfharm or harm to others as evidenced by endorsement of items 4 or 5 on the C-SSRS assessed prior to dosing on Day 1.
17. Received any of the following drugs listed, within 14 days or 5 half-lives (whichever islonger) before Day -1: Amiodarone, armodafinil, buproprion, Celecoxib, Cimetidine, Cinacalet, Ciproflaxin, Diphenhydramine, Duloxetine, Enoxacin, Escitalopram, Fluoxetine, Fluvoxamine, Gefitinib, Hydroxychloroquine, Methoxsalen, Mexiletine, Moclobemide, Paroxetine, Propafenone, Quinidine, Ranitidine, Ritonavir, Sertraline, Terbinafine, Thiabendazole, Ticlopidine, Voriconazole

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Peak and trough plasma concentrations following daily LUCEMYRA doses during clinic confinement | Day 1 (2, 3, 4, 5, 9 hours post dose), Days 2-4 (pre-dose and 4 hours post first daily dose), Taper Days 1-4 (pre-dose and 4 hours post first daily dose), Day of Discharge

SECONDARY OUTCOMES:
Estimation of apparent clearance and apparent volume of distribution for lofexidine and evaluation of possible covariates affecting PK | Day 1 post dose, Lucemyra fixed dosing days (4-8 days), Lucemyra Tapering days (4 days), discharge (1 day)
Treatment-emergent adverse events (TEAEs) | Day 1 post dose, Lucemyra fixed dosing days (4-8 days), Lucemyra Tapering days (4 days), safety monitoring (2.5 days), discharge (1 day), 30 day follow up
Vital signs: Heart Rate | Day -7 to -1, Dosing days (1 day up to 12 days), post last Lucemyra dose (Days 9 up to 14)
Vital Signs: Systolic blood pressure | Day -7 to -1, Dosing days (1 day up to 12 days), post last Lucemyra dose (Days 9 up to 14)
Vital Signs: Diastolic blood pressure | Day -7 to -1, Dosing days (1 day up to 12 days), post last Lucemyra dose (Days 9 up to 14)
Electrocardiograms (ECGs) QT Interval | Day -7 to -1, Day 3
Columbia-Suicide Severity Rating Scale (C-SSRS) | Day -7 to -1, Day 1, 2.5 days after last dose (discharge)
Number of participants with abnormal laboratory test results (hematology) | Day -7 to -1, 2.5 days after last dose (discharge)
  Safety laboratory assessments including blood tests for hematology will be performed.
Number of participants with abnormal laboratory test results (clinical chemistry) | Day -7 to -1, 2.5 days after last dose (discharge)
  Safety laboratory assessments including blood tests for clinical chemistry will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Mountain Manor Treatment Center, Baltimore, Maryland, United States